CLINICAL TRIAL: NCT04298710
Title: A Comparison Between the Effects of Different Muscle Groups on Blood Glucose Levels at the Postprandial Status in College Students
Brief Title: Effects of Arm Cycling and Leg Cycling on Postprandial Blood Glucose Levels in Healthy Persons
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research lab not accessible due to the pandemic.
Sponsor: Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Tongyu Ma, Assistant Professor of Health Sciences, Franklin Pierce University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CD02252020
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Hyperglycemia, Postprandial
MeSH Terms: conditions — Hyperglycemia | interventions — Sitting Position

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm Cycling (Experimental): Arm cycling on an arm crank ergometer for 20 minutes at light to moderate intensity. 30 minutes before the exercise, participants will consume 60g of carbohydrates mixed with plain water.
  Interventions: Behavioral: Arm Cycling
- Leg Cycling (Experimental): Leg cycling on a leg cycling ergometer for 20 minutes at light to moderate intensity. 30 minutes before the exercise, participants will consume 60g of carbohydrates mixed with plain water.
  Interventions: Behavioral: Leg Cycling
- Sitting (Placebo Comparator): Participants will remain seated after carbohydrates consumption.
  Interventions: Behavioral: Sitting

INTERVENTIONS:
Behavioral: Arm Cycling — 20 minutes of arm cycling exercise at light to moderate intensity.
  Arms: Arm Cycling
Behavioral: Leg Cycling — 20 minutes of leg cycling exercise at light to moderate intensity.
  Arms: Leg Cycling
Behavioral: Sitting — Remain seated for 20 minutes.
  Arms: Sitting

SUMMARY:
The literature has shown that exercise is effective in decreasing blood glucose levels. However, it remains less clear if there is any difference between muscle groups regarding the glucose-lowering effects of exercise. The purpose of this study is to examine the differences in blood-glucose level changes in response to exercise that involves different muscle groups.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy persons
* Age 18 years or above

Exclusion Criteria:

* Cardiovascular diseases
* Pulmonary diseases
* Metabolic diseases
* Other contraindications to exercise

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose levels | one hour after the carbohydrates intake

CONTACTS AND LOCATIONS:
Overall Officials: Tongyu Ma, Ph.D., Principal Investigator — Franklin Pierce University
Locations (1):
- Franklin Pierce University, Rindge, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No